CLINICAL TRIAL: NCT02878811
Title: China Patient-centered Evaluative Assessment of Cardiac Events (PEACE): Prospective Study of Patients With Heart Failure (HF)
Brief Title: China PEACE 5p-HF Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015BAI12B02-2
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure
Keywords: heart failure; prospective; cohort
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention: Samples With DNA Description: the investigators will collect plasma, serum, DNA, RNA, and urine at baseline and during follow-ups.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational study — This is a non-interventional study, patients receive their usual treatment as determined by the physician.

SUMMARY:
The investigators will consecutively recruit 5000 patients hospitalized for heart failure (HF) from 50 hospitals across China and follow them up for one year, describe treatment patterns during hospitalization and the follow-ups, examine patients recovery trajectory after HF, and identify targets for care quality improvement.

DETAILED DESCRIPTION:
This study will consecutively enroll patients with HF as the primary reason for hospitalization in 50 hospitals scattered all over China. Participants will be interviewed at baseline (i.e., during the index hospitalization for HF), and at 1, 6, and 12 months following hospital discharge. During the follow-up period, participants will be instructed to return to the hospital for interviews by site investigators. Telephone follow-ups will be conducted only when in-person interviews are not feasible.

At baseline, participants will be interviewed to collect detailed information about on demographics, socioeconomic status, cardiovascular risk factors, clinical characteristics, treatments, in-hospital outcomes, general and disease-specific quality of life, function and mental status; during the follow-ups, the investigators will collect information about clinical outcomes events, long-term treatments, function, quality of life, symptoms, and medical care during the recovery period.

The investigators will collect blood and urine samples during index hospitalization and the follow-ups.

This study will examine a series of factors that may affect patients' recovery after HF. Practical guidelines, quality evaluative system, and risk model will be established based on the findings, to improve patient outcomes in the future.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patients with heart failure as the primary reason for hospitalization, including both new-onset HF or decompensation of chronic HF
  2. Aged 18 years or above
* Exclusion Criteria:

  1. Patients who have enrolled in this study
  2. Patients who usually do not live in the city/county where the index hospital locates
  3. Patients who are unable to complete interviews due to severe conditions, mental illness, or communication difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with primary reason for admission of heart failure, aged 18 years or above
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1 year
  Major adverse cardiac events is defined as the composite of cardiovascular death, resuscitated sudden death, HF-related rehospitalization, myocardial infarction, stroke, and incident atrial fibrillation.

SECONDARY OUTCOMES:
Death | 1 year
  Cardiovascular death and non-cardiovascular death
Rehospitalization | 1 year
  HF-related and non HF-related
Resuscitated sudden death | 1 year
Myocardial infarction | 1 year
Stroke | 1 year
Incident atrial fibrillation | 1 year
Incident renal insufficiency | 1 year
Quality of life (EQ-5D) | 1 year
Quality of life for HF (KCCQ-12) | 1 year
Depression (PHQ-8) | 1 year
Stress (PSS-4) | 1 year
Anxiety (GAD-2) | 1 year
Function of cognition (Mini-cog) | 1 year

OTHER OUTCOMES:
Length of stay in hospital | 1 year
  For index hospitalization and accumulative during follow-up
Length of stay in ICU/CCU for index hospitalization | Duration of hospitalization, average of 10 days
Recurrent hospitalizations during study period | 1 year
Invasive procedures | 1 year
Prescription of proven therapies during hospitalization among ideal patients | Duration of hospitalization, average of 10 days
  Prescription of proven therapies (for HF medications, including dosage) during hospitalization among ideal patients (with indication and without contraindication)
Use of proven therapies during follow-up among ideal patients | 1 year
  Use of proven therapies (for HF medications, including dosage) during follow-up among ideal patients (with indication and without contraindication)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, PhD, Principal Investigator — China National Center for Cardiovascular Disease; Harlan M Krumholz, MD, SM, Principal Investigator — Yale University
Locations (1):
- Xinxiang Central Hospital, Xinxiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li J, Lei L, Wang W, Li Y, Yu Y, Pu B, Peng Y, Huo X, Zhang L. Patient-reported health status vs . N-terminal pro-B-type natriuretic peptide levels in patients with acute heart failure. Chin Med J (Engl). 2025 Nov 20;138(22):2955-2962. doi: 10.1097/CM9.0000000000003555. Epub 2025 Jul 22. PMID 40693625
- [Derived] Zhang L, Wang W, Peng Y, He G, Ji R, Lei L, Li J, Pu B, Liu Y, Yu Y, Zhang H. Associations of cumulative depressive symptoms within 1-year of discharge with subsequent mortality among patients hospitalized for acute heart failure: Findings from The China PEACE Prospective Heart Failure Study. J Affect Disord. 2024 Apr 15;351:299-308. doi: 10.1016/j.jad.2024.01.245. Epub 2024 Jan 28. PMID 38290578
- [Derived] Zhang L, He G, Huo X, Tian A, Ji R, Pu B, Peng Y. Long-Term Cumulative High-Sensitivity C-Reactive Protein and Mortality Among Patients With Acute Heart Failure. J Am Heart Assoc. 2023 Oct 3;12(19):e029386. doi: 10.1161/JAHA.123.029386. Epub 2023 Sep 30. PMID 37776214
- [Derived] Zhang L, Ji R, He G, Tian A, Huo X, Zheng Y, Qi L, Mi Y, Yan X, Wang B, Lei L, Li J, Liu J, Li J. Individual Trajectories of Health Status During the First Year of Discharge From Hospitalization for Heart Failure and Their Associations With Death in the Following Years. J Am Heart Assoc. 2023 Jul 18;12(14):e028782. doi: 10.1161/JAHA.122.028782. Epub 2023 Jul 8. PMID 37421271
- [Derived] Wang B, Lei L, Zhang H, Miao F, Zhang L, Tian A, Li J. Change in Depressive Symptoms During the First Month of Discharge and 1-Year Clinical Outcomes in Patients Hospitalized for Heart Failure. J Am Heart Assoc. 2022 Dec 20;11(24):e027438. doi: 10.1161/JAHA.122.027438. Epub 2022 Dec 14. PMID 36515248
- [Derived] Xing F, Zheng X, Zhang L, Hu S, Bai X, Hu D, Li B, Li J. Discharge heart rate and 1-year clinical outcomes in heart failure patients with atrial fibrillation. Chin Med J (Engl). 2022 Jan 5;135(1):52-62. doi: 10.1097/CM9.0000000000001768. PMID 34982055
- [Derived] Tian J, Zhao J, Zhang Q, Ren J, Han L, Li J, Zhang Y, Han Q. Assessment of chronic disease self-management in patients with chronic heart failure based on the MCID of patient-reported outcomes by the multilevel model. BMC Cardiovasc Disord. 2021 Jan 30;21(1):58. doi: 10.1186/s12872-021-01872-3. PMID 33516189
- [Derived] Huang X, Yu Y, Li X, Masoudi FA, Spertus JA, Yan X, Krumholz HM, Jiang L, Li J. The China Patient-centred Evaluative Assessment of Cardiac Events (PEACE) prospective heart failure study design. BMJ Open. 2019 Feb 19;9(2):e025144. doi: 10.1136/bmjopen-2018-025144. PMID 30782925